## Randomised Controlled Trial of Mechanochemical Ablation versus Cyanoacrylate Adhesive for the Treatment of Varicose Veins

## Statistical Analysis

Data were analysed using SPSS version 27 and Stata version 26 on an intention-to-treat basis. Normality of the distribution of the data was assessed using visual inspection, Kolmogorov-Smirnov and Shapiro-Wilk tests. Normally distributed continuous data were presented as mean and standard deviation and analysed using parametric tests; otherwise presented as median and interquartile range and analysed using non-parametric tests. Accordingly, either one-way repeated measures analysis of variance or related samples of Friedman's Two-Way Analysis of Variance were used for paired data. Bonferroni correction was used where appropriate. Chi-squared tests were applied for categorical data and reported as frequencies and proportions (as percentages). When we designed the study, the critical level of significance was set at 0.05 (5%). However, as interim analyses were carried out one year from the beginning of recruitment, 42,43 the alpha spending function of Lan and DeMets approaches 44,45 was used to control the number of Type I errors.